CLINICAL TRIAL: NCT05764356
Title: Imapct of bioMarkers on Pharmacodynamics and Bleeding Risk of Direct Oral AntiCoagulants and Ticagrelor Study II (IMPACT 2)
Brief Title: Imapct of bioMarkers on Pharmacodynamics and Bleeding Risk of Direct Oral AntiCoagulants and Ticagrelor Study II
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Cui Yimin, Prof., Peking University First Hospital
Other Study IDs: 2022CR67
Record Dates: First submitted 2023-02-16; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Novel Oral Anticoagulants; NOACs; Rivaroxaban; Apixaban; Edoxaban; Dabigatran; Ticagrelor; Pharmacodynamics; Pharmacogenomics; RNA Profile; Bleeding; Biomarker
MeSH Terms: conditions — Hemorrhage | interventions — Platelet Count; Leukocyte Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Novel oral anticoagulants cohort
  Interventions: Genetic: Detection of genotype and RNA profile in platelet and white blood cell; Other: Indicators test related to coagulation function
- Ticagrelor cohort
  Interventions: Genetic: Detection of genotype and RNA profile in platelet and white blood cell; Other: Indicators test related to platelet function

INTERVENTIONS:
Genetic: Detection of genotype and RNA profile in platelet and white blood cell — Detection of genotype by next generation sequencing Detection of RNA profile in platelet and white blood cell by RNA sequencing
Other: Indicators test related to coagulation function — Indicators test including prothrombin time (PT), activated partial thrombin time (APTT), thrombin time (TT), diluted TT (dTT), snake vein enzyme coagulation time (ECT), anti-XA or IIa activity, etc.
  Groups: Novel oral anticoagulants cohort
Other: Indicators test related to platelet function — Indicators test related to platelet function. Platelet reactivity was measured by VASP. Platelet aggregation rate was measured by turbidimetric method. Platelet and fibrinolytic function were measured by thrombologram, etc.
  Groups: Ticagrelor cohort

SUMMARY:
Individual differences in drug efficacy and adverse reactions are common in the clinical application of drugs. Individual differences are caused by many factors, among which genetic factors account for more than 20%. Novel oral anticoagulant drugs (NOACs, including rivaroxaban, apixaban, edoxaban, dabigatran, etc.) and novel antiplatelet drug ticagrelor have the advantages of convenient use and no need for monitoring. But novel oral antithrombotic drugs also increase the risk of bleeding, and there is currently a lack of effective antagonists when antithrombosis is excessive or emergency surgery is required. At present, there are few studies on the causes of individual differences in novel antithrombotic drugs, and there is a lack of predictable biomarkers or drug genotypes, especially in China. Therefore, on the basis of previous studies on NOACs and ticagrelor individualized medication cohorts, this study plans to establish a validation cohort for novel antithrombotic drugs bleeding related biomarkers, conduct multi-omics testing and long-term follow-up, and explore markers related to pharmacodynamics of antithrombotic drugs, adverse bleeding reactions and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

(I) Chinese Patients taking NOACs

* In accordance with anticoagulation indications of NOACs, include prevention of thrombosis in non valvular atrial fibrillation, prevention and treatment of deep vein thrombosis / pulmonary embolism and prevention of thrombosis after knee / hip replacement;
* More than 18 years of age, male or female;
* Never received NOACs in a month and intend to take NOACs or have received NOACs for more than one week continuously;
* sign informed consent.

(II) Chinese Patients taking ticagrelor

* With diagnosis of acute coronary syndrome (ACS), included unstable angina, non ST segment elevation myocardial infarction and ST segment elevation myocardial infarction;
* More than 18 years of age, male or female;
* Never received ticagrelor in a month and intend to take ticagrelor or have received ticagrelor for more than one week continuously#
* sign informed consent.

Exclusion Criteria:

* With history of immunodeficiency disease, including positive HIV index;
* Positive Hepatitis B surface antigen (HBsAg) and HCV index;
* Combined therapy of CYP3A4 strong inhibitors and P-gp inhibitors (e.g., systemic pyrrole antifungal agents such as ketoconazole, itraconazole, voriconazole and posaconazole; human immunodeficiency virus (HIV) - protease inhibitors such as ritonavir), CYP3A4 strong inducers and P-gp inducers (e.g., rifampicin, phenytoin, phenobarbital, carbamazepine, St. John's Wort, etc.) in 14 days before treatment with NOACs;
* Severe liver dysfunction and abnormal renal function;
* Include contraindications of antithrombosis, such as hypersensitivity, active bleeding, moderate or severe liver disease, previous history of intracranial hemorrhage, gastrointestinal hemorrhage in the past 6 months and major operation within 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese Patients taking NOACs or ticagrelor#In accordance with anticoagulation indications of NOACs or with diagnosis of acute coronary syndrome (ACS)# received NOACs or ticagrelor in a month and intend to take NOACs or ticagrelor, or have received NOACs or ticagrelor for more than one week continuously#1000 patients for each cohort (NOACs or ticagrelor).
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of new bleeding events | Within 1 month after enrollment
  During the observation time, record the incidence of new bleeding events after NOACs(rivaroxaban, apixaban, edoxaban, dabigatran) or ticagrelor administration by telephone and out-patient clinic, including subcutaneous bleeding, gingival bleeding, gastrointestinal bleeding, intracranial hemorrhage, etc.
Incidence of new bleeding events | From 1 month to 6 months after enrollment
  During the observation time, record the incidence of new 'bleeding events after NOACs(rivaroxaban, apixaban, edoxaban, dabigatran) or ticagrelor administration by telephone and out-patient clinic, including subcutaneous bleeding, gingival bleeding, gastrointestinal bleeding, intracranial hemorrhage, etc.
Incidence of new bleeding events | From 6 months to 1 year after enrollment
  During the observation time, record the incidence of new bleeding events after NOACs(rivaroxaban, apixaban, edoxaban, dabigatran) or ticagrelor administration by telephone and out-patient clinic, including subcutaneous bleeding, gingival bleeding, gastrointestinal bleeding, intracranial hemorrhage, etc.
Incidence of new bleeding events | From 1 year to 2 years after enrollment
  During the observation time, record the incidence of new bleeding events after NOACs(rivaroxaban, apixaban, edoxaban, dabigatran) or ticagrelor administration by telephone and out-patient clinic, including subcutaneous bleeding, gingival bleeding, gastrointestinal bleeding, intracranial hemorrhage, etc.
Incidence of new major cardiovascular events and all-cause death | Within 1 month after enrollment
  During the observation time, record the new incidence of major cardiovascular events (MACEs) and all-cause death after NOACs(rivaroxaban, apixaban, edoxaban, dabigatran) or ticagrelor administration by telephone and out-patient clinic. MACEs including cardiac death, myocardial infarction (MI), stroke or transient cerebral thrombus (TIA), ischemic-driven coronary revascularization(PCI, CABG, thrombolysis, etc.), etc.
Incidence of new major cardiovascular events and all-cause death | From 1 month to 6 months after enrollment
  During the observation time, record the new incidence of major cardiovascular events (MACEs) and all-cause death after NOACs(rivaroxaban, apixaban, edoxaban, dabigatran) or ticagrelor administration by telephone and out-patient clinic. MACEs including cardiac death, myocardial infarction (MI), stroke or transient cerebral thrombus (TIA), ischemic-driven coronary revascularization(PCI, CABG, thrombolysis, etc.), etc.
Incidence of new major cardiovascular events and all-cause death | From 6 months to 1 year after enrollment
  During the observation time, record the new incidence of major cardiovascular events (MACEs) and all-cause death after NOACs(rivaroxaban, apixaban, edoxaban, dabigatran) or ticagrelor administration by telephone and out-patient clinic. MACEs including cardiac death, myocardial infarction (MI), stroke or transient cerebral thrombus (TIA), ischemic-driven coronary revascularization(PCI, CABG, thrombolysis, etc.), etc.
Incidence of new major cardiovascular events and all-cause death | From 1 year to 2 years after enrollment
  During the observation time, record the new incidence of major cardiovascular events (MACEs) and all-cause death after NOACs(rivaroxaban, apixaban, edoxaban, dabigatran) or ticagrelor administration by telephone and out-patient clinic. MACEs including cardiac death, myocardial infarction (MI), stroke or transient cerebral thrombus (TIA), ischemic-driven coronary revascularization(PCI, CABG, thrombolysis, etc.), etc.
Incidence of new thromboembolic events | Within 1 month after enrollment
  During the observation time, record the incidence of new thromboembolic events after NOACs(rivaroxaban, apixaban, edoxaban, dabigatran) or ticagrelor administration by telephone and out-patient clinic, including stroke or TIA, systemic embolism (SE), deep vein thrombosis (DVT), pulmonary embolism, left auricular thrombus, stent thrombosis, stent stenosis and stent endothelial hyperplasiastent, etc.
Incidence of new thromboembolic events | From 1 month to 6 months after enrollment
  During the observation time, record the incidence of new thromboembolic events after NOACs(rivaroxaban, apixaban, edoxaban, dabigatran) or ticagrelor administration by telephone and out-patient clinic, including stroke or TIA, systemic embolism (SE), deep vein thrombosis (DVT), pulmonary embolism, left auricular thrombus, stent thrombosis, stent stenosis and stent endothelial hyperplasiastent, etc.
Incidence of new thromboembolic events | From 6 months to 1 year after enrollment
  During the observation time, record the incidence of new thromboembolic events after NOACs(rivaroxaban, apixaban, edoxaban, dabigatran) or ticagrelor administration by telephone and out-patient clinic, including stroke or TIA, systemic embolism (SE), deep vein thrombosis (DVT), pulmonary embolism, left auricular thrombus, stent thrombosis, stent stenosis and stent endothelial hyperplasiastent, etc.
Incidence of new thromboembolic events | From 1 year to 2 years after enrollment
  During the observation time, record the incidence of new thromboembolic events after NOACs(rivaroxaban, apixaban, edoxaban, dabigatran) or ticagrelor administration by telephone and out-patient clinic, including stroke or TIA, systemic embolism (SE), deep vein thrombosis (DVT), pulmonary embolism, left auricular thrombus, stent thrombosis, stent stenosis and stent endothelial hyperplasiastent, etc.

SECONDARY OUTCOMES:
Genotype detected by next generation sequencing | Through study completion, collection only once
  Collect blood specimen before NOACs administration, then detect genotype of NOACs by next generation sequencing.
Expression level of RNA in platelet and white blood cell | NOACs: Once each before administration, before and after administration at stable concentration (at least 48h for rivaroxaban, 72h for apixaban or edoxaban). Ticagrelor: Once before administration and once after stable concentration (at least 48h).
  Before and after NOACs or ticagrelor administration, detect the expression level of RNA in platelet and white blood cell .
Anticoagulantion activity evaluation (for NOACs only) | Once each before administration, before and after administration at stable concentration (at least 48h for rivaroxaban, 72h for apixaban or edoxaban) .
  Before and after NOACs administration, record anti-factor Xa activity(for rivaroxaban, apixaban, edoxaban) or anti-factor IIa activity (for dabigatran only) detected by blood coagulation tests.
Platelet reactivity evaluation (for Ticagrelor only) | Once before administration and once after stable concentration.
  Before and after ticagrelor administration, record PRI detected by one or more following methods: 1)LTA; 2)VASP ELISA test; 3)TEG.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Anhui Provincial Hospital#The First Affiliated Hospital Of USTC#, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital Of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The 7th People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital FuDan University, Shanghai, Shanghai Municipality